CLINICAL TRIAL: NCT07214324
Title: Integrative Multi-omics Analysis to Predict Monoclonal Gammopathies Clinical Evolution
Acronym: PNRR-2022-1237
Status: Active, not recruiting | Type: Observational
Sponsor: Azienda USL Reggio Emilia - IRCCS (Other Government)
Collaborators: European Union Next Generation (Unknown); Ministero della Salute, Italy (Other)
Responsible Party: Sponsor
Other Study IDs: 849/2022/TESS/IRCCSRE
Record Dates: First submitted 2025-10-02; First posted 2025-10-09 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-10

CONDITIONS: Monoclonal Gammopathy of Undetermined Significance (MGUS); Smoldering Multiple Myeloma (SMM); Multiple Myeloma (MM)
Keywords: plasma cells; multi-omics; biomarkers; bone marrow microenvironment; microbiome
MeSH Terms: conditions — Monoclonal Gammopathy of Undetermined Significance; Smoldering Multiple Myeloma; Multiple Myeloma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Malignant plasma cells were purified from bone marrow mononuclear cells, and genomic DNA was extracted for subsequent genomic analyses.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- MGUS, SMM and MM patients: Patients with monoclonal gammopathy of undeterminated significance, smoldering multiple myeloma, or multiple myeloma
  Interventions: Other: Collection of biological material
- Healthy volunteers: Patients with a clinical and radiological diagnosis of osteoarthritis who undergo endo or arthro-prosthesis surgery
  Interventions: Other: Collection of biological material

INTERVENTIONS:
Other: Collection of biological material — For MGUS, SMM and MM patients, biological material (bone marrow aspirate, bone marrow biopsy, peripheral blood) consists exclusively of left-over samples obtained during routine diagnostic procedures and clinical practice management of their disease.
  For healthy volunteers, biological material includes waste bone tissue obtained during orthopedic surgery (endo- or arthro-prosthesis) and peripheral blood collected for research purposes.
  Both cohort of patient will be asked to donate gingival crevicular fluid (GCF) (this is a non-invasive procedure with no associated risks).

SUMMARY:
This prospective, multicenter, observational study aims to identify molecular and immunological markers associated with disease progression in patients with monoclonal gammopathy of undetermined significance (MGUS) and smoldering multiple myeloma (SMM). By integrating genomic, transcriptomic, immunophenotypic, and oral microbiome analyses, the study seeks to characterize the biological mechanisms underlying the transition to symptomatic multiple myeloma (MM). The study also includes in vitro modeling to investigate bone damage and immune dysfunction. Healthy volunteers (HV) undergoing joint replacement surgery for osteoarthritis will serve as controls. The ultimate goal is to improve early risk stratification and support future preventive strategies through a multi-omics approach. There is a pressing need for new strategies to identify high-risk individuals based on biological rather than purely clinical parameters. This study proposes an integrative, multi-omics approach to investigate the transition from MGUS/SMM to MM. By analyzing the immunome and oral microbiome alongside molecular profiling, the goal is to identify reliable biomarkers of progression. The resulting insights could be enable more accurate risk stratification and guide the design of future preventive clinical trials aimed at delaying or halting disease evolution.

DETAILED DESCRIPTION:
Multiple myeloma (MM) is a hematologic malignancy characterized by the clonal proliferation of antibody-secreting plasma cells in the bone marrow. It accounts for approximately 10% of all blood cancers, with an incidence of 3-5per 100.000 individuals in Westen countries. MM is an incurable disease that leads to severe bone destruction and fractures due to the abnormal interaction between malignant plasma cells and the bone marrow microenvironment. Although new therapies have improved survival, MM remains a complex and genetically heterogeneous disease. Genomic instability is a hallmark of MM and includes both chromosomal abnormalities and gene mutations. Tumors may presenta s hyperdiploid - with multiple trisomies - or non-hyperdiploid, often involving translocations at the immunoglobulin heavy chain locus (IGH). These genetic differences impact prognosis. Additional recurrent alterations, such as deletions (13q, 17q), gains (1q), and mutations in genes like KRAS, NRAS, TP53, and BRAF, further illustrate the disease's biological diversity. Molecular profiling techniques, such as RNA sequencing and gene expression arrays, have identified gene expression patterns that correlate with prognosis, though only a few are currently used in clinical practice. MM is consistently preceded by two asymptomatic precursor conditions: monoclonal gammopathy of undetermined significance (MGUS) and smoldering multiple myeloma (SMM). These conditions are prevalent in older adults and share many molecular features with symptomatic MM, yet only a small fraction of cases progress annually - about 1% for MGUS and 10% for SMM. Disease evolution appears to depend not only on intrinsic genetic changes but also on interactions with the bone marrow microenvironment, which includes stromal cells, dendritic cells, T cells (especially Th17), NK cells and myeloid-derived suppressors cells. Immune dysfunction, antigen presentation defects, expansion of immunosuppressive cells, and high levels of inhibitory cytokines contribute to the emergence of an immunosuppressive niche that enables myeloma cells to escape immune surveillance and progress. Immunomodulatory drugs (ImiDs) and monoclonal antibodies, which can reactivate immune responses, are therefore central to treatment strategies. Recent evidence also suggests a link between the microbiota and disease progression. In experimental models, alterations in gut microbiota have been shown to affect immune responses, influencing disease onset. Currently available prognostic tools mainly reflect tumor burden rather than underlying biology. As such, they fail to accurately predict disease progression.

ELIGIBILITY:
Inclusion Criteria:

* Age >18 years
* Male or female patients
* Histologically confirmed diagnosis of MGUS, SMM, or MM according to ESMO 2021 guidelines
* Willing and able to provide written informed consent

HEALTHY VOLUNTEERS (HV)

* Age >60 years
* Diagnosis of osteoarthritis (OA)
* Scheduled for hospitalization for surgical treatment of OA (endoprosthesis or arthroplasty)
* Willing and able to provide written informed consent

Exclusion Criteria:

* Patients:

  * Active current infection
  * Autoimmune disease
  * Women of childbearing potential unable to exclude pregnancy
  * Use of high-dose corticosteroids within the past 7 days, potentially affecting immunome composition

Healthy Volunteers:

* Prior joint surgery or severe joint deformity
* Recent trauma, osteonecrosis, or OA caused by prior/current joint infection
* Metabolic disorders
* Previous or current cancer diagnosis
* Autoimmune diseases (e.g., rheumatoid arthritis)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: patients with MGUS, SMM, or MM (with or without bone lytic lesions), as well as patient with osteoarthritis undergoing joint surgery (endoprosthesis or artroplasty) (Healty Volunteers)
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2023-01-01 (Actual); Primary Completion 2025-08-12 (Actual); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Bone marrow and peripheral blood immunophenotypic characterization | up to 24 months
  Multiparametric flow cytometry of bone marrow CD138- cells and peripheral blood mononuclear cells (PBMCs) to define immune subsets and to assess alterations associated with monoclonal gammopathies progression.
Genomic and transcriptomic profiling of plasma cell | Up to 24 months
  Next-generation sequencing (NGS) analysis of bone marrow CD138+ plasma cells, including targeted 14-gene mutation panels, copy number alterations by ultra-low-pass whole genome sequencing, RNA sequencing, and single-cell transcriptomics to identify molecular signatures of disease evolution.
Single-cell and spatial transcriptomic analyses | up to 24 months
  Single-cell RNAseq, antibody-based sequencing (ABseq), TCR sequencing, and spatial transcriptomics on bone marrow biopsies to characterize clonal heterogeneity, cell-cell interactions, and microenvironmental influences during progression from MGUS/SMM to Multiple Myeloma.

SECONDARY OUTCOMES:
Evaluation of oral microbiome composition | up to 24, months
  Sequencing-based profiling (16S rRNA) of DNA extracted from gingival crevicular fluid (GCF) samples of patients and healthy volunteers to investigate oral microbiome dysbiosis and its association with immune dysfunction and disease progression.
Functional validation of genetic profiles in osteolytic disease | 24 months
  Use of CRISPR-Cas9 screening in myeloma cell lines and dynamic 3D co-culture models (osteoblasts, osteoclasts, immune and stromal cells) to evaluate the role of specific molecular pathways in osteolytic lesion development and immune impairment.

CONTACTS AND LOCATIONS:
Overall Officials: Antonino Neri, MD, PhD, Study Chair — Azienda USL - IRCCS di Reggio Emilia
Locations (4):
- Italy (4):
  - Istituto Ortopedico Rizzoli IRCCS, Bologna
  - UO Ematologia Azienda Ospedaliero-Universitaria "Policlinico Rodolico San Marco", Catania
  - UOC di Ematologia, Dipartimento di Oncologia, AOU Policlinico "Paolo Giaccone", Palermo
  - S.C Ematologia - Azienda USL IRCCS di Reggio Emilia, Reggio Emilia

REFERENCES:
- [Background] Rossi M, Altomare E, Botta C, Gallo Cantafio ME, Sarvide S, Caracciolo D, Riillo C, Gaspari M, Taverna D, Conforti F, Critelli P, Bertucci B, Iannone M, Polera N, Scumaci D, Arbitrio M, Amodio N, Di Martino MT, Paiva B, Tagliaferri P, Tassone P. miR-21 antagonism abrogates Th17 tumor promoting functions in multiple myeloma. Leukemia. 2021 Mar;35(3):823-834. doi: 10.1038/s41375-020-0947-1. Epub 2020 Jul 6. PMID 32632096
- [Background] Leone P, Solimando AG, Malerba E, Fasano R, Buonavoglia A, Pappagallo F, De Re V, Argentiero A, Silvestris N, Vacca A, Racanelli V. Actors on the Scene: Immune Cells in the Myeloma Niche. Front Oncol. 2020 Oct 29;10:599098. doi: 10.3389/fonc.2020.599098. eCollection 2020. PMID 33194767
- [Background] Bolli N, Maura F, Minvielle S, Gloznik D, Szalat R, Fullam A, Martincorena I, Dawson KJ, Samur MK, Zamora J, Tarpey P, Davies H, Fulciniti M, Shammas MA, Tai YT, Magrangeas F, Moreau P, Corradini P, Anderson K, Alexandrov L, Wedge DC, Avet-Loiseau H, Campbell P, Munshi N. Genomic patterns of progression in smoldering multiple myeloma. Nat Commun. 2018 Aug 22;9(1):3363. doi: 10.1038/s41467-018-05058-y. PMID 30135448
- [Background] Ziccheddu B, Da Via MC, Lionetti M, Maeda A, Morlupi S, Dugo M, Todoerti K, Oliva S, D'Agostino M, Corradini P, Landgren O, Iorio F, Pettine L, Pompa A, Manzoni M, Baldini L, Neri A, Maura F, Bolli N. Functional Impact of Genomic Complexity on the Transcriptome of Multiple Myeloma. Clin Cancer Res. 2021 Dec 1;27(23):6479-6490. doi: 10.1158/1078-0432.CCR-20-4366. Epub 2021 Sep 15. PMID 34526359
- [Background] Robiou du Pont S, Cleynen A, Fontan C, Attal M, Munshi N, Corre J, Avet-Loiseau H. Genomics of Multiple Myeloma. J Clin Oncol. 2017 Mar 20;35(9):963-967. doi: 10.1200/JCO.2016.70.6705. Epub 2017 Feb 13. PMID 28297630
- [Background] Morgan GJ, Walker BA, Davies FE. The genetic architecture of multiple myeloma. Nat Rev Cancer. 2012 Apr 12;12(5):335-48. doi: 10.1038/nrc3257. PMID 22495321
- [Background] Palumbo A, Anderson K. Multiple myeloma. N Engl J Med. 2011 Mar 17;364(11):1046-60. doi: 10.1056/NEJMra1011442. No abstract available. PMID 21410373